CLINICAL TRIAL: NCT01918917
Title: Phase 4 Study of Intra-articular Dexmedetomidine Adding to Levobupivacaine for Postoperative Analgesia in Arthroscopic Knee Surgery
Brief Title: Adding Intra-articular Dexmedetomidine to Levobupivacaine for Postoperative Analgesia in Arthroscopic Knee Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Ulgey, Assisstant Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011/329; 2011/329 (Registry Identifier: Erciyes University Ethic Committe)
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Pain
Keywords: Arthroscopic knee surgery; Dexmedetomidine; Analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Levobupivacaine; Dexmedetomidine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levobupivacaine (Active Comparator): Intraarticular 19 ml 0.5% levobupivacaine and 1 ml 0.9% sodium chloride administered. postoperative morphine administered for analgesia
  Interventions: Drug: Levobupivacaine; Drug: Dexmedetomidine; Drug: Morphine
- Dexmedetomidine (Active Comparator): Intraarticular 19 ml 0.5% levobupivacaine and 1 ml (100 mcg/ml) dexmedetomidine administered, postoperative morphine used for analgesia
  Interventions: Drug: Dexmedetomidine; Drug: Morphine

INTERVENTIONS:
Drug: Levobupivacaine — intraarticular
  Other Names: chirocaine 0.5%
  Arms: Levobupivacaine
Drug: Dexmedetomidine — intraarticular 1 ml (100 mcg)
  Other Names: precedex, 100mcg/ml
Drug: Morphine — intravenously, patient-controlled analgesia
  Other Names: morphine HCL, 10 mg

SUMMARY:
The purpose of this study to search efficacy of intra-articular dexmedetomidine addition to levobupivacaine for postoperative analgesia in arthroscopic knee surgery.

DETAILED DESCRIPTION:
Patients between 18-65 years and with American Society of Anesthesiologists' (ASA) Physical Status class I-II, who were scheduled for arthroscopic knee surgery, were enrolled in a randomised comparative clinical trial. Blinding or masking began in the preoperative holding unit. Exclusion criteria were psychiatric illness, younger than 18 yo, who has analgesic treatment before the surgery and known hypersensitivity to relevant drugs. All patients received a standard anaesthetic protocol; ECG, heart rate, non-invasive blood pressure, oxygen saturation and temperature were monitored. After preoxygenation, general anaesthesia was induced with sodium pentothal 4 to 7 mg/kg, 1 mcg/kg fentanyl and neuromuscular block was achieved with rocuronium 0.5 mg/kg and trachea was intubated. Anesthesia was maintained with desflurane 6% and 50% oxygen in the medical air.

Randomised patients were achieved dexmedetomidine and levobupivacaine or levobupivacaine intra-articularly 10 minutes before medical tourniquet deaerated.

Postoperative analgesia was maintained with morphine in patient-controlled analgesia. Patients postoperative VAS values and analgesic consumptions were recorded in postoperative 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 yo
* scheduled for arthroscopic knee surgery

Exclusion Criteria:

* younger than 18 yo
* known allergy relevant drugs
* contraindication for general anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Analgesic consumption | up to 48 hours

SECONDARY OUTCOMES:
blood pressure | before deaerate the medical tourniquet, after deaerate the tourniquet, postoperative 0, 30, 60, 90, 120 minutes ,in the PACU, 4, 6, 12, 24, 48 hours
heart rate | before deaerate the medical tourniquet, after deaerate the tourniquet, postoperative 0, 30, 60, 90, 120 minutes ,in the PACU, 4, 6, 12, 24, 48 hours
Visual Analog Scale-rest | postoperative 0, 30, 60, 90, 120 minutes in the PACU, 4, 6, 12, 24, 48 hours
Visual Analog Scale-movement | postoperative 0, 30, 60, 90, 120 minutes ,in the PACU, 4, 6, 12, 24, 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Resul Altuntas, MD, Principal Investigator — TC Erciyes University; Ayse Ulgey, Ast Prof, Study Director — TC Erciyes University